CLINICAL TRIAL: NCT04347902
Title: Intravenous Lipid Emulsions and Liver Function in Adult Chronic Intestinal Failure Patients: New Results After 5 Years.
Brief Title: Lipid Emulsions and Liver Function - Results After 5 Years.
Acronym: 5ylipids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the General Surgery Unit, Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lipids-5 year
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Liver Failure; Parenteral Nutrition-Related Hepatitis
MeSH Terms: conditions — Liver Failure | interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PN with SMOFLipid (Experimental): Parenteral nutrition with MCT/LCT/olive oil/fish oil (SMOFLipid, Fresenius Kabi, Germany, SMOF group)
  Interventions: Drug: Intravenous Lipid Emulsion
- PN with Olive oil (Active Comparator): Parenteral nutrition with Olive oil/LCT 80:20 (ClinOleic, Baxter Healthcare, USA, OO group)
  Interventions: Drug: Intravenous Lipid Emulsion
- PN with MCT/LCT (Active Comparator): Parenteral nutrition with - Medium/long-chain triglycerides 50:50 (Lipofundin, B Braun Germany, MCT/LCT group)
  Interventions: Drug: Intravenous Lipid Emulsion

INTERVENTIONS:
Drug: Intravenous Lipid Emulsion — Various types of intravenous lipids

SUMMARY:
Intravenous lipid emulsion (ILE) is an essential component of parenteral nutrition (PN), but also one of the key risk factors for development of intestinal failure associated liver disease (IFALD). The aim of the study was to analyse the influence of ILEs on liver function during long term PN.

DETAILED DESCRIPTION:
Intravenous lipid emulsion (ILE) is an essential component of parenteral nutrition (PN), but also one of the key risk factors for development of intestinal failure associated liver disease (IFALD). Despite of many commercially available ILEs with hypothetically different impact on liver, a direct comparison of them has never been performed. Therefore the aim of the study was to analyse the influence of ILEs on liver function during long term PN. Ths study is a continuation of the previous trial, NCT03044639.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age,
* chronic intestinal failure on PN including lipids,
* metabolic stability (the absence of pathological laboratory resulting in the change of PN regime for at least one month)
* ability to tolerate up to 1.0 g lipids/kg body weight per day as a part of PN

Exclusion Criteria:

* preexisting liver dysfunction (an elevation of SGOT, SGTP, total bilirubin, GGTP, alkaline phosphatase of more than 3 times x normal value),
* patients with a history of cancer and anti-cancer treatment within the last 5 years,
* severe hyperlipidemia,
* severe coagulopathy,
* severe renal insufficiency,
* acute thromboembolic events,
* positive test for HIV, Hepatitis B or C (from medical history),
* known or suspected drug or alcohol abuse,
* participation in another interventional clinical trial in parallel or within three months prior to the start of this clinical trial,
* for women with childbearing potential (i.e. females who are not chemically or surgically sterile or females who are not postmenopausal) or women of childbearing potential tested positive on standard pregnancy test (urine dipstick) or/and lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Liver disfunction | 5 years
  Liver tests results during parenteral nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, PhD, Principal Investigator — Stanley Dudrick's Memorial Hospital
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klek S, Szczepanek K, Scislo L, Walewska E, Pietka M, Pisarska M, Pedziwiatr M. Intravenous lipid emulsions and liver function in adult chronic intestinal failure patients: results from a randomized clinical trial. Nutrition. 2018 Nov;55-56:45-50. doi: 10.1016/j.nut.2018.03.008. Epub 2018 Mar 22. PMID 29960156